CLINICAL TRIAL: NCT00986479
Title: An Investigation of the Antidepressant Effects of an NMDA Antagonist in Treatment-Resistant Major Depression
Brief Title: This is a Study to Determine the Antidepressant Effects of AZD6765
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6702C00015; NCT00995111 (obsolete NCT alias)
Record Dates: First submitted 2009-09-24; First posted 2009-09-30 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Treatment Resistant Major Depressive Disorder
Keywords: Patients
MeSH Terms: interventions — AZD6765

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD6765 (150 mg) / Placebo (Experimental): Patients randomized to receive a single intravenous (iv) infusion of AZD6765 (150 mg) over 60 minutes during the first period, followed by a 7-day drug-free period, followed by a single iv infusion of placebo (saline solution) over 60 minutes during the second period.
  Interventions: Drug: AZD6765
- Placebo / AZD6765 (150 mg) (Placebo Comparator): Patients randomized to receive a single intravenous (iv) infusion of placebo (saline solution) over 60 minutes during the first period, followed by a 7-day drug-free period, followed by a single iv infusion of AZD6765 (150 mg) over 60 minutes during the second period.
  Interventions: Drug: Placebo to AZD6765

INTERVENTIONS:
Drug: AZD6765 — Single IV infusion of 150 mg AZD6765.
  Arms: AZD6765 (150 mg) / Placebo
Drug: Placebo to AZD6765 — Single IV infusion of Placebo to AZD6765
  Arms: Placebo / AZD6765 (150 mg)

SUMMARY:
The purpose of this study is to determine the antidepressant effects of AZD6765 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Major Depressive Disorder, currently depressed without psychotic features
* Females must be of non-childbearing potential.

Exclusion Criteria:

* Treatment with Clozapine or ECT within 3 months prior to study
* Current or past history of psychotic features or a diagnosis of schizophrenia or any other psychotic disorder as defined in the DSM-IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, MD, Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- Research Site, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Lepow L, Luckenbaugh DA, Park L, Henter ID, Zarate CA Jr. Case series: Antidepressant effects of low-affinity and low-trapping NMDA receptor antagonists did not predict response to ketamine in seven subjects. J Psychiatr Res. 2017 Mar;86:55-57. doi: 10.1016/j.jpsychires.2016.10.023. Epub 2016 Nov 22. No abstract available. PMID 27914292
- [Derived] Zarate CA Jr, Mathews D, Ibrahim L, Chaves JF, Marquardt C, Ukoh I, Jolkovsky L, Brutsche NE, Smith MA, Luckenbaugh DA. A randomized trial of a low-trapping nonselective N-methyl-D-aspartate channel blocker in major depression. Biol Psychiatry. 2013 Aug 15;74(4):257-64. doi: 10.1016/j.biopsych.2012.10.019. Epub 2012 Dec 1. PMID 23206319
- See also: D6702C00015 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=213&filename=D6702C00015_Clinical_Study_Report_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 patients were enrolled. Of these, 22 patients were randomized to either: (1) AZD6765 (150 mg) followed by placebo or (2) placebo followed by AZD6765 (150 mg) in a crossover study design. A total of 20 patients completed both treatment periods of the study.
Pre-assignment Details: Screening for eligibility and washout of restricted medications.
Groups:
- AZD6765 (150 mg): Patients randomized to receive a single intravenous (iv) infusion of AZD6765 (150 mg) over 60 minutes during the first period, followed by a 7-day drug-free period, followed by a single iv infusion of placebo (saline solution) over 60 minutes during the second period.
- Placebo: Patients randomized to receive a single intravenous (iv) infusion of placebo (saline solution) over 60 minutes during the first period, followed by a 7-day drug-free period, followed by a single iv infusion of AZD6765 (150 mg) over 60 minutes during the second period.
Period: Period 1
Arm/Group | AZD6765 (150 mg) | Placebo
Started | 12 | 10
Completed | 10 | 10
Not Completed | 2 | 0
Not completed — Improved mood | 1 | 0
Not completed — Administrative reasons | 1 | 0
Period: Period 2
Arm/Group | AZD6765 (150 mg) | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AZD6765 (150 mg)/ Placebo: Patients randomized to receive a single intravenous (iv) infusion of AZD6765 (150 mg) over 60 minutes during the first period, followed by a 7-day drug-free period, followed by a single iv infusion of placebo (saline solution) over 60 minutes during the second period.
- Placebo/AZD6765 (150 mg): Patients randomized to receive a single intravenous (iv) infusion of placebo (saline solution) over 60 minutes during the first period, followed by a 7-day drug-free period, followed by a single iv infusion of AZD6765 (150 mg) over 60 minutes during the second period.
- Total: Total of all reporting groups
Arm/Group | AZD6765 (150 mg)/ Placebo | Placebo/AZD6765 (150 mg) | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (10.9) | 52.4 (10.5) | 51.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Total Score.
Description: Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item instrument used for the evaluation of depressive symptoms. Each item is rated on a scale of 0 to 6 (with higher scores indicating more severe depression). The individual item scores are added together to form a total score, ranging between 0 and 60. 0 is considered the best score, 60 the worst.
Time Frame: 60 minutes (min) prior to dosing (baseline); and 60 min, 80 min, 110 min, 230 min, 1 day, 2 days, 3 days and 7 days following dosing.
Population: ITT population including all randomized patients who were given study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  60 minutes | 26.881 (1.262) | 28.618 (1.314)
  80 minutes | 25.381 (1.262) | 29.718 (1.314)
  110 minutes | 25.835 (1.262) | 29.818 (1.314)
  230 minutes | 26.517 (1.262) | 29.418 (1.314)
  Day 1 | 27.654 (1.262) | 29.118 (1.314)
  Day 2 | 29.161 (1.288) | 31.368 (1.314)
  Day 3 | 30.732 (1.288) | 30.368 (1.314)
  Day 7 | 31.447 (1.288) | 31.222 (1.342)

2. Secondary Outcome: The Number of Participants With Montgomery-Asberg Depression Rating Scale (MADRS) Total Score Less Than 10 (MADRS Remission).
Description: Remission defined as a Montgomery-Asberg Depression Rating Scale (MADRS) total score <10. MADRS is a 10-item instrument used for the evaluation of depressive symptoms. Each item is rated on a scale of 0 to 6 (with higher scores indicating more severe depression). The individual item scores are added together to form a total score, ranging between 0 and 60. 0 is considered the best score, 60 the worst.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Number; unit: Participants
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Participants
  60 minutes | 2 | 1
  80 minutes | 4 | 0
  110 minutes | 4 | 0
  230 minutes | 2 | 0
  Day 1 | 2 | 0
  Day 2 | 1 | 0
  Day 3 | 1 | 0
  Day 7 | 1 | 0

3. Secondary Outcome: The Number of Participants With at Least 50% Reduction in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score (MADRS Response).
Description: Response defined as a >= 50% reduction from baseline in MADRS total score. MADRS is a 10-item instrument used for the evaluation of depressive symptoms. Each item is rated on a scale of 0 to 6 (with higher scores indicating more severe depression). The individual item scores are added together to form a total score, ranging between 0 and 60. 0 is considered the best score, 60 the worst.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Number; unit: Participants
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Participants
  60 minutes | 5 | 3
  80 minutes | 6 | 1
  110 minutes | 4 | 0
  230 minutes | 4 | 1
  Day 1 | 3 | 0
  Day 2 | 1 | 0
  Day 3 | 1 | 0
  Day 7 | 1 | 0

4. Secondary Outcome: Scale for Suicide Ideation (SSI) Total Score.
Description: Scale for Suicide Ideation (SSI) is a 19-item scale designed to quantify the intensity of current conscious suicide ideation. Each item is rated on a scale of 0 to 2 (with higher scores indicating greater suicidal ideation). The individual item scores are added together to form a total score, ranging between 0 and 38. 0 is considered the best outcome, 38 the worst.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  60 minutes | 0.955 (0.326) | 0.939 (0.330)
  80 minutes | 1.137 (0.326) | 1.039 (0.330)
  110 minutes | 1.137 (0.326) | 0.989 (0.330)
  230 minutes | 0.864 (0.326) | 0.939 (0.330)
  Day 1 | 1.364 (0.326) | 1.539 (0.330)
  Day 2 | 1.236 (0.328) | 1.189 (0.330)
  Day 3 | 1.379 (0.328) | 1.226 (0.332)
  Day 7 | 1.379 (0.328) | 1.507 (0.332)

5. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A) Total Score.
Description: Hamilton Anxiety Rating Scale (HAM-A) is used as a rating measure of anxiety severity. The scale consists of 14 items. Each item is rated on a scale of 0 to 4. The HAM-A total score is the sum of the 14 items and the score ranges from 0 to 56. 0 is considered the best outcome, 56 the worst.
Time Frame: 60 minutes (min) prior to dosing (baseline); and 230 min, 1 day, 2 days, 3 days and 7 days following dosing.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  230 minutes | 16.211 (1.181) | 17.160 (1.207)
  Day 1 | 16.666 (1.181) | 17.675 (1.198)
  Day 2 | 16.817 (1.190) | 18.125 (1.198)
  Day 3 | 17.055 (1.190) | 18.525 (1.198)
  Day 7 | 18.817 (1.190) | 19.631 (1.207)

6. Secondary Outcome: Hamilton Depression Rating Scale-17 Item (HDRS) Total Score
Description: Hamilton Depression Rating Scale-17 item (HDRS) is a scale that assesses depressive symptoms. HDRS consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher scores indicate more severe depression.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  60 minutes | 15.930 (0.977) | 17.389 (1.008)
  80 minutes | 14.975 (0.977) | 17.739 (1.008)
  110 minutes | 15.475 (0.977) | 18.039 (1.008)
  230 minutes | 16.112 (0.977) | 17.339 (1.008)
  Day 1 | 16.748 (0.977) | 17.639 (1.008)
  Day 2 | 16.732 (0.977) | 19.289 (1.008)
  Day 3 | 17.732 (0.977) | 19.039 (1.008)
  Day 7 | 18.160 (0.991) | 19.438 (1.024)

7. Secondary Outcome: Visual Analogue Scale (VAS) Depressed Score
Description: The Visual Analog Scale (VAS) Depressed is a 0 to 100-mm self-administered scale where patients rate their mood between "extreme sad" (0-mm) and "extreme happy" (100-mm), with a median "normal" point.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Scores on a scale
  60 minutes | 55.614 (6.137) | 60.562 (6.197)
  80 minutes | 58.614 (6.137) | 57.662 (6.197)
  110 minutes | 60.750 (6.137) | 59.062 (6.197)
  230 minutes | 55.614 (6.137) | 61.212 (6.197)
  Day 1 | 62.160 (6.137) | 64.762 (6.197)
  Day 2 | 65.753 (6.166) | 63.262 (6.197)
  Day 3 | 66.896 (6.166) | 63.312 (6.197)
  Day 7 | 68.467 (6.166) | 65.576 (6.264)

8. Secondary Outcome: Clinician-Administered Dissociative States Scale (CADSS) Score.
Description: Clinician- Administered Dissociative States Scale (CADSS) is a clinician-administered measure of perceptual, behavioral, and attentional alterations occurring during dissociative experiences. This scale involves a 23 questions and each is rated from 0 (not at all) to 4 (extremely). The total score is sum of the 23 items and range from 0 to 92 - best is 0 and worst is 92.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  60 minutes | 4.104 (0.900) | 1.997 (0.921)
  80 minutes | 3.324 (0.909) | 2.297 (0.921)
  110 minutes | 2.831 (0.900) | 2.047 (0.921)
  230 minutes | 1.240 (0.900) | 1.497 (0.921)
  Day 1 | 1.013 (0.900) | 1.147 (0.921)
  Day 2 | 1.360 (0.910) | 1.397 (0.921)
  Day 3 | 1.456 (0.910) | 1.447 (0.921)
  Day 7 | 1.313 (0.910) | 1.212 (0.932)

9. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) Score.
Description: The Brief Psychiatric Rating Scale (BPRS) is a 18-item scale which measures symptoms and behaviors that are characteristic of schizophrenia. Each item is rated from 1 to 7 with higher score indicating greater severity. The total score is the sum of the 18 items, resulting in a range of scores from 18-126.
  18 is considered to be the best outcome, 126 the worst.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  60 minutes | 32.191 (1.271) | 32.896 (1.314)
  80 minutes | 30.237 (1.271) | 33.496 (1.314)
  110 minutes | 30.555 (1.271) | 33.696 (1.314)
  230 minutes | 30.737 (1.271) | 31.772 (1.314)
  Day 1 | 33.418 (1.271) | 33.596 (1.314)
  Day 2 | 32.882 (1.291) | 34.496 (1.314)
  Day 3 | 34.168 (1.291) | 33.046 (1.314)
  Day 7 | 35.739 (1.291) | 34.428 (1.335)

10. Secondary Outcome: Beck Depression Inventory (BDI) Score.
Description: Beck Depression Inventory (BDI) is a 21-question instrument for measuring the severity of depression. Each question has a set of at least four possible answer choices, ranging in intensity. A value of 0 to 3 is assigned for each answer and the total score is computed. Higher total scores indicate more severe depressive symptoms.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  60 minutes | 21.081 (2.524) | 22.886 (2.538)
  80 minutes | 22.217 (2.524) | 23.122 (2.546)
  110 minutes | 21.535 (2.524) | 23.586 (2.538)
  230 minutes | 21.126 (2.524) | 23.686 (2.538)
  Day 1 | 22.444 (2.524) | 22.936 (2.538)
  Day 2 | 22.923 (2.531) | 24.586 (2.538)
  Day 3 | 23.494 (2.531) | 23.786 (2.538)
  Day 7 | 24.447 (2.531) | 24.070 (2.546)

11. Secondary Outcome: Young Mania Rating Scale (YMRS) Score.
Description: Young Mania Rating Scale (YMRS) consists of 11 items, rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe) or from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60. 0 is considered to be the best outcome, 60 the worst.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  60 minutes | 4.294 (0.412) | 3.626 (0.427)
  80 minutes | 3.748 (0.412) | 3.526 (0.427)
  110 minutes | 3.475 (0.412) | 3.526 (0.427)
  230 minutes | 3.748 (0.412) | 3.526 (0.427)
  Day 1 | 3.748 (0.412) | 3.326 (0.427)
  Day 2 | 3.699 (0.419) | 3.676 (0.427)
  Day 3 | 4.270 (0.419) | 3.476 (0.427)
  Day 7 | 4.366 (0.419) | 4.339 (0.435)

12. Secondary Outcome: Visual Analogue Scale (VAS) Anxious Score.
Description: The Visual Analog Scale (VAS) Anxious is a 0 to 100-mm self-administered scale where patients rate their mood between "extreme sad" (0-mm) and "extreme happy" (100-mm), with a median "normal" point.
Time Frame: as for outcome 1
Population: ITT population including all randomized patients who were given study treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  60 minutes | 43.898 (7.415) | 41.929 (7.479)
  80 minutes | 44.216 (7.415) | 44.079 (7.479)
  110 minutes | 42.853 (7.415) | 44.729 (7.479)
  230 minutes | 44.580 (7.415) | 46.029 (7.479)
  Day 1 | 44.989 (7.415) | 47.229 (7.479)
  Day 2 | 44.718 (7.447) | 50.479 (7.479)
  Day 3 | 42.623 (7.447) | 48.279 (7.479)
  Day 7 | 50.147 (7.447) | 56.595 (7.551)

13. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS) Positive Score.
Description: Brief Psychiatric Rating Scale (BPRS) Positive is a 4-item scale which measures positive symptoms of schizophrenia (conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content). Each item is rated from 1 to 7 with higher score indicating greater severity. The total score is the sum of the 4 items, resulting in a range of scores from 4-28.
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZD6765 (150 mg) | Placebo
Number analyzed (Participants) | 22 | 20
Units on a scale
  60 minutes | 9.433 (0.264) | 8.946 (0.274)
  80 minutes | 8.751 (0.264) | 8.996 (0.274)
  110 minutes | 8.660 (0.264) | 8.996 (0.274)
  230 minutes | 8.751 (0.264) | 8.666 (0.279)
  Day 1 | 9.114 (0.264) | 9.296 (0.274)
  Day 2 | 9.118 (0.269) | 9.296 (0.274)
  Day 3 | 9.118 (0.269) | 9.446 (0.274)
  Day 7 | 9.356 (0.269) | 9.338 (0.279)

ADVERSE EVENTS:
Arm/Group | AZD6765 (150 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 21/22 | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD6765 (150 mg) (N=22) | Placebo (N=20)
Bradycardia (Cardiac disorders) | 1 | 1
Hypertension (Vascular disorders) | 8 | 5
Hypotension (Vascular disorders) | 3 | 1
Tachycardia (Cardiac disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 2
Vision blurred (Eye disorders) | 2 | 1
Eye irritation (Eye disorders) | 1 | 1
Decreased apetite (Metabolism and nutrition disorders) | 9 | 5
Increased apetite (Metabolism and nutrition disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 2
Flatulence (Gastrointestinal disorders) | 2 | 3
Thirst (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 3
Abdominal discomfort (Gastrointestinal disorders) | 6 | 5
Faeces discoloured (Gastrointestinal disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Weight increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 1
Libido increased (Nervous system disorders) | 1 | 0
Felt faint (Nervous system disorders) | 10 | 3
Headache (Nervous system disorders) | 2 | 4
Dental care (Surgical and medical procedures) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 5 | 3
Gingival disorder (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 1
Oedema (General disorders) | 1 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Tic (Psychiatric disorders) | 1 | 1
Tremor (Nervous system disorders) | 3 | 4
Malignant dysphagia (Gastrointestinal disorders) | 1 | 1
Influenza (Infections and infestations) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 3
Disturbance in attention (Psychiatric disorders) | 10 | 6
Confusional state (Psychiatric disorders) | 6 | 1
Depression (Psychiatric disorders) | 4 | 1
Initial insomnia (Psychiatric disorders) | 7 | 8
Somnolence (Psychiatric disorders) | 15 | 12
Terminal insomnia (Psychiatric disorders) | 6 | 7
Hallucination (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 10 | 11
Irritability (Nervous system disorders) | 10 | 8
Memory impairment (Nervous system disorders) | 5 | 5
Hypokinesia (Nervous system disorders) | 7 | 6
Psychomotor activity (Psychiatric disorders) | 5 | 4
Dysarthria (Nervous system disorders) | 3 | 1
Suicidal behaviour (Nervous system disorders) | 1 | 0
Suicidal ideation (Nervous system disorders) | 2 | 3
Fatigue (General disorders) | 6 | 5
Skin irritation (Skin and subcutaneous tissue disorders) | 3 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 1
Surgery (Surgical and medical procedures) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 3 | 2
Body temperature decreased (Investigations) | 5 | 4
Dissociation (Psychiatric disorders) | 3 | 2
Euphoric mood (Nervous system disorders) | 3 | 0
Social avoindant behaviour (Psychiatric disorders) | 4 | 3
Abnormal behaviour (Nervous system disorders) | 8 | 3
Feeling abnormal (Psychiatric disorders) | 5 | 3
Body temperature increased (Investigations) | 5 | 3
Energy increased (General disorders) | 5 | 1
Hypoaesthesia (Nervous system disorders) | 6 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Fear of falling (Psychiatric disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 6 | 2
Visual impairment (Eye disorders) | 3 | 1
Abnormal dreams (Nervous system disorders) | 3 | 5
False Sensation (Psychiatric disorders) | 9 | 6
Dizziness (Nervous system disorders) | 10 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No